CLINICAL TRIAL: NCT04735679
Title: Multi-omic Longitudinal Characterization of Pulmonary Microbiome in Cystic Fibrosis Patients
Brief Title: Characterization of Pulmonary Microbiome in Cystic Fibrosis Patients
Acronym: SPutOM-CF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0053
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Cystic Fibrosis
Keywords: MICROBIOLOGY; MULTI-OMIC; SPUTUM; PULMONARY MICROBIOTA; CYSTIC FIBROSIS; COHORT; ANTIBIOTHERAPY
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The composition and role of the pulmonary microbiota is not yet well described in cystic fibrosis patients.

The objective of our longitudinal follow-up of primary colonised patients is to show the presence of a link between the composition of the microbiota and the effectiveness of antibiotic therapy.

All patients followed at the Montpellier CF center will be asked to participate in this cohort. All patients have a regular follow-up every 1 to 6 months and will be asked at each visit to keep their sputum sample in excess of the analyses requested for their follow-up

DETAILED DESCRIPTION:
The composition and role of the pulmonary microbiota is not yet well described in cystic fibrosis patients.

According to our hypothesis, the lung microbiota shapes the lung environment of cystic fibrosis patients and modifies the effectiveness of antibiotic treatments and the course of the disease. The objective of our longitudinal follow-up of primary colonised patients is to show the presence of a link between the composition of the microbiota and the effectiveness of antibiotic therapy. Finally, the management of first colonisations could justify the characterisation of the microbiota in order to develop innovative diagnostic tests for the follow-up of patients suffering from cystic fibrosis and possibly the identification of new therapeutic agents based on the microbiota.

All patients followed at the Montpellier CF centre will be asked to participate in this cohort. All patients have a regular follow-up every 1 to 6 months and will be asked at each visit to keep their sputum sample in excess of the analyses requested for their follow-up.

ELIGIBILITY:
Inclusion criteria:

- Cystic fibrosis patient

Exclusion criteria

- Refusal to participate in this research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic fibrosis patients
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
to determine a characterisation of the microorganisms of the lung microbiota | 1 day
  to characterise the microorganisms of the lung microbiota and their interspecific interactions by taxonomic and functional analyses.
to determine a ink between the Composition of the microbiota | 1 day
  To demonstrate the relationship between the composition of the microbiota and the evolution of the disease Defines the effectiveness of anti-inflammatory biotherapy in patients with cystic fibrosis
to determine a Effectiveness of antibiotic therapy | 1 day
  To identify abiotic conditions that may contribute to the gap between the efficacy of antibiotics in vitro and in vivo.
  Show that the microbiota plays a role in the effectiveness of antibiotic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael CHIRON, PU-PH, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC